CLINICAL TRIAL: NCT05134051
Title: Microcirculatory Status After Intravascular Lithotripsy
Acronym: MARVEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiac Research Institute BV (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/066
Record Dates: First submitted 2021-10-31; First posted 2021-11-24 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Chronic Coronary Insufficiency; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: The MARVEL Pilot STUDY is an investigator-initiated, multicenter, single-arm, open-label, assessing the microcirculation after IVL and PCI in severe calcific stenoses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): single arm intervention with IVL in calcified de novo coronary stenoses with indication of plaque modification technique during PCI
  Interventions: Device: Shockwave® Intravascular Lithotripsy System (Shockwave Medical Inc)

INTERVENTIONS:
Device: Shockwave® Intravascular Lithotripsy System (Shockwave Medical Inc) — IVL is a novel balloon catheter-based device that utilises pulsatile mechanical energy to disrupt calcified lesions. IVL differs from other types of lithotripsy with respect to depth of penetration. It is a single-use, sterile, disposable balloon catheter. The emitters convert electrical energy into transient acoustic circumferential pressure pulses that disrupt both superficial and deep calcium within plaque. The balloon catheter is connected to the generator, which is programmed to deliver the specified dosage of pulses. The IVL balloon, sized 1:1 to the reference artery ratio, is inflated low pressure (4 atm) with 10 pulses of ultrasound energy of 10s delivered per balloon. The procedure is repeated to provide a minimum of 20 pulses in the target lesion, with interval deflation to allow distal perfusion. Each catheter can emit a max of 80 pulses at a rate of one pulse per second. If the lesion exceeds the 12mm balloon length, the balloon can be repositioned and the IVL repeated.

SUMMARY:
Due to differences in the mechanism of action, intravascular lithotripsy is likely to cause less distal embolization and microcirculatory dysfunction during plaque preparation. This may also translate into lower periprocedural myocardial infarction rates. Thus, this exploratory study aims to evaluate the microcirculatory function after the use of Shockwave® intravascular lithotripsy.

DETAILED DESCRIPTION:
Patients with stable coronary artery disease or stabilized acute coronary syndromes with severely calcified de novo coronary stenoses with indication of plaque modification technique during PCI.

Due to differences in the mechanism of action, intravascular lithotripsy is likely to cause less distal embolization and microcirculatory dysfunction during plaque preparation. This may also translate into lower periprocedural myocardial infarction rates.

To perform the invasive physiology assessment an intracoronary pressure and temperature sensor-tipped guidewire is used to measure distal coronary pressure and to derive thermodilution curves. For the calculation of IMR three thermodilution curves can be obtained from a hand-held, 3-ml rapid (<0.25s) injection of room temperature saline at baseline and during maximal hyperemia. Mean transit time (Tmn) at baseline and during maximal hyperemia is derived from the thermodilution curves. Simultaneous recordings of mean aortic pressure (guiding catheter, Pa) and mean distal coronary pressure (distal pressure sensor, Pd) is also obtained at baseline and during maximal hyperemia. The IMR is then calculated using the following equation: IMR = PaxTmn[(Pd-Pw)/(Pa-Pw)], where Pw is the coronary wedge pressure. Pw will be measured as the distal coronary pressure (from the distal pressure and temperature sensor) during complete balloon occlusion of the vessel obtained during PCI.

The aim of the present study is to investigate the protective effect of IVL (Shockwave© Medical) on the coronary microcirculatory during PCI in calcific coronary stenosis, compared to RA.

ELIGIBILITY:
Inclusion Criteria:

* Angiographic inclusion criteria

  * Severely calcified stenoses
  * Vessels with RVD between 2.5 - 4.0 mm
  * TIMI flow 3

Exclusion Criteria:

* Angiographic exclusion criteria

  * Concomitant use of rotational atherectomy
  * Severe vessel tortuosity
  * Stenosis un-crossable with a balloon/guidewire
  * Concomitant conditions
  * Contraindication for adenosine administration.
  * Hemodynamic or electrical instability.
  * Active liver disease or hepatic dysfunction, defined as AST or ALT > 3 times the ULN.
  * Severe renal dysfunction, defined as an eGFR <30 mL/min/1.73 m2, unless the patient is in renal support therapy.
* Other exclusion criteria

  * Unable to provide written informed consent (IC)
  * Known pregnancy or breast-feeding at time of inclusion; pre-menopausal women, unless sterilized, must take an effective method of birth control up to 15 weeks after the end of treatment with IP
  * Prior myocardial infarction subtended to the PCI target vessel.
  * Akinesia or dyskinesia in myocardial segments in the distribution area of the PCI target vessel.
  * Severe systolic dysfunction defined as left ventricular ejection fraction < 35%.
  * Patent arterial or venous surgical graft supplying the PCI target vessel.
  * Previous TIMI flow < 1 before guidewire crossing.
  * Patient not eligible for drug-eluting stent treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Index of Microcirculatory Resistance (IMR) after IVL | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Post-PCI FFR after IVL | through study completion, an average of 1 year
Rate of periprocedural myocardial infarction | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Collet, Principal Investigator — Cardiovascular Center OLV Aalst
Locations (1):
- Hospital San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No